CLINICAL TRIAL: NCT06504212
Title: Reliability and Validity Of A Mobile Applicatıon in the Evaluation of Elbow Joint Position Sense
Brief Title: Validity and Reliability of a New Mobile Application
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gülfem Ezgi ÖZALTIN, PhD, physiotherapist, Principal Investigator, Inonu University
Other Study IDs: 2024/5554(2)
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Proprioception
Keywords: mobile application; validity; reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
In this study, we aimed to study the validity and reliability of the Angle Meter, a Smartphone application for elbow joint position sense.

DETAILED DESCRIPTION:
The validity and reliability of the elbow joint position sense with the mobile application will be evaluated with the angle meter. This application works on phones with the IOS operating system. The validity and reliability of the Angle Meter will be evaluated by comparing it with a small universal goniometer for measuring elbow range of motion. The elbows of healthy subjects will be photographed at 3 different angles in the open and kinetic chain position. The elbow photo of healthy individuals measured with the Angle meter will be evaluated simultaneously but independently with the Angle meter by 2 different evaluators. The measurements will be repeated after 3 days. It will be noted that each picture is sufficient, i.e. there is no obvious perspective error.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being healthy
* Agreeing to participate in the study

Exclusion Criteria:

* Those who have had upper extremity surgery within the last year
* Those with neurological, orthopedic, rheumatic or cardiovascular problems affecting the neck, shoulder, elbow, hand and wrist
* Those with central and peripheral nervous system involvement Having pain anywhere in the body

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2024-07-12 (Estimated); Primary Completion 2024-10-12 (Estimated); Study Completion 2024-11-12 (Estimated)

PRIMARY OUTCOMES:
universal goniometer | [Time Frame: 3 days]
  Joint position sense measurement with universal goniometer .
mobile application | [Time Frame: 3 days]
  The elbows will be photographed in 3 different angles, in open and kinetic chain position. The elbow photograph of healthy individuals measured with the Angle meter will be evaluated simultaneously but independently with the Angle meter by 2 different evaluators.

CONTACTS AND LOCATIONS:
Overall Officials: dilan demirtas karaoba, Study Chair — Inonu University; havva adli, Study Chair — Inonu University; burcu talu, Study Chair — Inonu University
Locations (1):
- Gulfem Ezgi, Malatya, Inonu University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No